CLINICAL TRIAL: NCT05539157
Title: A Phase 1 Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of JCXH-211 Intratumoral Injection in Patients With Malignant Solid Tumors
Brief Title: Study to Evaluate JCXH-211 as Monotherapy in Patients With Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Immorna Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-JCXH-211-001
Record Dates: First submitted 2022-08-30; First posted 2022-09-14 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Cutaneous Tumor; Malignant Solid Tumor
Keywords: Tumor; Intratumoral injection
MeSH Terms: conditions — Skin Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a:Dose escalation (Experimental): JCXH-211 will be delivered by intratumoral injection in 3 stages:
  Single administration stage A single administration of JCXH-211 administered to cutaneous or subcutaneous lesions in escalating doses.
  Multiple administration stage Up to 3 doses of JCXH-211 administered to a cutaneous or subcutaneous lesion in escalating doses. Assigned dose to be determined on the data from the single administration arm.
  Visceral administration stage JCXH-211 administered to a visceral lesion in escalating doses. Assigned dose to be determined on the data from the single and multiple administration arms.
  Interventions: Drug: JCXH-211
- Phase 1b:Dose expansion (Experimental): JCXH-211 will be delivered by intratumoral injection. The dose to be used will be determined after review of the data from Phase 1a.
  Interventions: Drug: JCXH-211

INTERVENTIONS:
Drug: JCXH-211 — JCXH-211 administered once every 28 days

SUMMARY:
A Phase 1 Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of JCXH-211 Intratumoral Injection in Patients with Malignant Solid Tumors

DETAILED DESCRIPTION:
The main purpose of this study is to find out how safe and tolerable the study drug, JCXH-211, is and also how well it works in people with malignant solid tumors. The study drug JCXH-211, is an immunotherapy drug. This means that it aims to work by boosting immune system's response to tumors, to help fight against the growth of the cancer cells. The study has 2 main phases: Phase 1a and Phase 1b. Phase 1a has 3 stages, Single administration stage, Multiple administration stage and Visceral stage. Phase 1b will not start until all the data collected in Phase 1a has been completed and reviewed to check that it is safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

All of the following conditions should be met at screening:

* Male or female patients 18-75
* Patients with malignant solid tumors that have been diagnosed by pathology and/or cytology
* Patients who have progressed on or who cannot tolerate available therapies or for whom curative therapy does not exist
* Patients with at least one non-injected measurable tumor lesion per RECIST v1.1
* Patients with lesions suitable for intratumoral injection (the lesion length is at least 10 mm and not exceeding 80 mm)
* Patients enrolled in the single and multiple administration stages of Phase 1a must agree to provide pre- and post-treatment tumor biopsy tissues
* Patients must have adequate organ and marrow functions
* Patients with treated brain metastases are eligible if meeting protocol's requirement
* Patients must be ≥ 4 weeks beyond treatment with any chemotherapy (6 weeks for nitrosoureas or mitomycin C), hormonal, biological, targeted agents, other investigational therapy or radiotherapy

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

* Patients who have received prior IL-12 either alone or as part of a treatment regimen
* Patients who have received prior therapy with an immuno-oncology agent and were discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (irAE)
* Patients requiring therapeutic doses of anticoagulation
* Patients with tumors that impinge on major airways, blood vessels, or nerve bundles
* Patients with a history of autoimmune disease that has the possibility of recurrence or active autoimmune disease that requires immunosuppressive medications
* Patients who had a major surgical procedure within 4 weeks prior to the first dose of study treatment
* Current or prior use of immunosuppressive medication within 2 weeks prior to the first dose of study treatment
* Patient with history of solid organ or allogenic bone marrow transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | Day 1 to Day 29
  Dose limiting toxicity, evaluated in the single administration stage of Phase 1a, which will be used to determine the MTD and to determine dose escalation
Incidence of adverse events (Safety and Tolerability) | From consent to 30 days after the last dose of study drug
  Safety and tolerability as determined by the incidence of adverse events (AEs), including severe AEs and serious AEs (SAEs)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 12 months
  Objective response rate is defined as the proportion of patients that achieve a complete response (CR) or partial response (PR) during the study participation.
Duration of response (DOR) | Up to 12 months following first reported response
  Duration of response is defined as the time from the first assessment of tumor as CR or PR to the first assessment as progressive disease or death from any cause.
Time to response (TTR) | Up to 12 months from the start of study therapy
  Time to response is defined as the time from Day 1 until the first documentation of objective response (CR or PR).
Disease control rate (DCR) | Up to 12 months
  Disease control rate is defined as the proportion of patients with CR or PR or stable disease (SD) with the DOR ≥ 12 weeks observed from Day 1 to disease progression.
Progression-free survival (PFS) | Up to 12 months
  Progression-free survival is defined as the time from Day 1 to disease progression or death from any cause, whichever occurs earlier.
Overall survival (OS) | Up to 24 months
  Overall survival is defined as the time from Day 1 until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No